CLINICAL TRIAL: NCT03955146
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Pamrevlumab in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Zephyrus I: Evaluation of Efficacy and Safety of Pamrevlumab in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study did not meet its primary endpoint.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-091
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis, IPF, Idiopathic Interstitial Pneumonia, Interstitial Lung Disease, Lung Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — pamrevlumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Main Study Cohort: Pamrevlumab (Experimental): Participants will receive pamrevlumab 30 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion every 3 weeks for up to 48 weeks in the DB period.
  Interventions: Drug: Pamrevlumab
- Main Study Cohort: Placebo (Placebo Comparator): Participants will receive placebo matching to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks in the DB period.
  Interventions: Drug: Placebo
- Japan Extension Cohort: Pamrevlumab (Experimental): Participants will receive pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
  Interventions: Drug: Pamrevlumab
- Japan Extension Cohort: Placebo (Placebo Comparator): Participants will receive placebo matching to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks.
  Interventions: Drug: Placebo
- OLE Period: Pamrevlumab/Pamrevlumab (Experimental): Participants who receive pamrevlumab in the DB period will continue to receive the same dose of pamrevlumab for up to 48 weeks in the OLE period or until pamrevlumab is commercially available for the indication of IPF, or the sponsor decides to end the OLE period, whichever occurrs first.
  Interventions: Drug: Pamrevlumab
- OLE Period: Placebo/Pamrevlumab (Experimental): Participants who receive placebo matching to pamrevlumab in the DB period, will receive pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the OLE period or until pamrevlumab is commercially available for the indication of IPF, or the sponsor decides to end the OLE period, whichever occurrs first.
  Interventions: Drug: Pamrevlumab

INTERVENTIONS:
Drug: Pamrevlumab — Pamrevlumab will be administered per dose and schedule specified in the arm description.
  Other Names: FG-3019
  Arms: Japan Extension Cohort: Pamrevlumab; Main Study Cohort: Pamrevlumab; OLE Period: Pamrevlumab/Pamrevlumab; OLE Period: Placebo/Pamrevlumab
Drug: Placebo — Placebo matching to pamrevlumab will be administered per schedule specified in the arm description.
  Arms: Japan Extension Cohort: Placebo; Main Study Cohort: Placebo

SUMMARY:
This is a Phase 3 trial to evaluate the efficacy and safety of 30 milligrams (mg)/kilogram (kg) intravenous (IV) infusions of pamrevlumab administered every 3 weeks as compared to placebo in participants with IPF.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multi-center trial to evaluate the efficacy and safety of pamrevlumab in participants with IPF.

Participants who are not being treated with approved IPF therapies (that is, nintedanib or pirfenidone) may be eligible for screening. Examples of reasons participants may not be treated with approved IPF therapies include but are not limited to:

* Intolerant or not responsive to approved IPF therapies
* Ineligible to receive these therapies
* Participant voluntarily declines to receive approved IPF therapies after being fully informed of the potential benefits/risks

NOTE: No participant should discontinue an approved IPF therapy for the purpose of enrolling in this study.

The study consists of the following study periods:

* Main (double blind, placebo-controlled) phase:

  * Screening period: Up to 6 weeks
  * Treatment period: 48 weeks
* Optional, open-label extension (OLE) phase of pamrevlumab:

  o Access to pamrevlumab will be available until the last participant completes 48 weeks of treatment in the OLE phase, or pamrevlumab is commercially available for the indication of IPF, or the Sponsor decides to end the OLE phase, whichever occurs first.
* Follow-up period/final safety assessments:

  * 28 days after last dose
  * 60 days after last dose: follow-up phone call, for a final safety assessment

During the treatment period, co-administration of an approved IPF therapy (that is, pirfenidone or nintedanib) is acceptable if clinically indicated in the Investigator's opinion, provided that the Investigator assesses the potential risks/benefits of combining approved IPF therapies with blinded study treatment.

Participants who discontinue study treatment for any reason should be encouraged to remain in the study and be followed for all study visits and assessments.

Participants who complete the Week 48 visit of the main study (regardless of the number of study drug infusions received) will be eligible to participate in the optional OLE phase of the study that offers continuing access to pamrevlumab regardless of randomization assignment in the main study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of IPF as defined by American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japan Radiological Society (JRS)/Latin American Thoracic Association (ALAT) guidelines within the past 7 years prior to study participation.
2. High-resolution computed tomography (HRCT) scan at screening, with ≥10% to <50% parenchymal fibrosis (reticulation) and <25% honeycombing.
3. FVCpp value >45% and <95% at screening and Day 1 (prior to randomization).
4. Diffusing capacity of the lungs for carbon monoxide (DLCO) percent predicted and corrected by hemoglobin (Hb) value ≥25% and ≤90% at screening (determined locally).
5. Not currently receiving treatment for IPF with an approved therapy (that is, pirfenidone or nintedanib) for any reason, including prior intolerance or lack of response to an approved IPF therapy, or choice to forego treatment with an approved IPF therapy after a full discussion with the Investigator regarding risks/benefits of such therapy.

Key Exclusion Criteria:

1. Previous exposure to pamrevlumab.
2. Evidence of significant obstructive lung disease.
3. Female participants who are pregnant or nursing.
4. Smoking within 3 months of screening and/or unwilling to avoid smoking throughout the study.
5. Interstitial lung disease other than IPF.
6. Sustained improvement in the severity of IPF during the 12 months prior to screening.
7. History of other types of respiratory diseases including diseases or disorders of the airways, lung parenchyma, pleural space, mediastinum, diaphragm, or chest wall.
8. Medical conditions (for example, myocardial infarction [MI]/stroke within the past 6 month), or logistical challenges that in the opinion of the Investigator preclude the participant's adequate participation in the study.
9. Acute IPF exacerbation during screening or randomization.
10. Use of any investigational drugs or unapproved therapies, or participation in any clinical trial with an investigational new drug within 30 days prior to screening. Or use of approved IPF therapies (that is, pirfenidone or nintedanib) within 1 week prior to screening.
11. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies, or to any component of the excipient.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (125):
- United States (60):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - Norton Thoracic Institute, Phoenix, Arizona
  - Pulmonary Associates, PA - Research, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - J&L Research, Conway, Arkansas
  - Loma Linda University Health, Loma Linda, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - St. Francis Medical Center, Clearwater, Florida
  - University of Florida Pulmonary, Critical Care & Sleep Medicine Division, Gainesville, Florida
  - University of Florida Health, Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Pulmonary Disease Specialist, PA d/b/a, PDS Research, Kissimmee, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare, Inc., Austell, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University of Chicago, Maywood, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Pulmonary Health Physicians, PC, Liverpool, New York
  - Pulmonix, LLC, Greensboro, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Legacy Research Institute, Portland, Oregon
  - The Oregon Clinic, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Comprehensive Lung and Sleep Center, Hendersonville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Pulmonary Sleep, Allergy and Asthma Associates, Cypress, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Utah Health, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - Fundacion Respirar - Centro Médico Dra. De Salvo, Ciudad Autonoma de Buenos Aires (caba), Buenos Aires
  - Centro de Investigacion Metabolica 'CINME', Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Consultorios Medicos. Organización del Buen Ayre. SRL, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico de Enfermedades Respiratorias, Florida, Buenos Aires
  - Centro Platense en Investigaciones Respiratorias, La Plata, Buenos Aires
  - Instituto ave Pulmo Fundacion enfisema, Mar del Plata, Buenos Aires
  - Respira Salud Clinica Integral, Godoy Cruz, Mendoza Province
  - INSARES, Mendoza, Mendoza Province
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
- Australia (6):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Health Services Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Chile (4):
  - Centro Investigacion del Maule CIM, Talca, Maule Region
  - Instituto Nacional del Torax, Santiago, Santiago Metropolitan
  - CIMER, Santiago, Santiago Metropolitan
  - M y F estudios clinicos, Santiago, Santiago Metropolitan
- China (22):
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - BeiJing Chao-Yang Hospital,Capital medical university, Beijing, Beijing Municipality
  - China-Japan friendship hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen people's hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Provincial chest hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital，Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - People's Hospital of Inner Mongolia Autonomous Region, Hohhot, Inner Mongolia
  - The second hospital of Dalian medical university, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Huaxi Hospital of Sichuan University., Chengdu, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
- Hong Kong (2):
  - Queen Mary Hospital, Central
  - Tuen Mun Hospital, Hong Kong
- Russia (10):
  - Regional Clinical Hospital #3, Chelyabinsk
  - Kazan State Medical University based on Republican Clinical Hospital, Kazan'
  - Clinical Hospital #3, Kemerovo
  - Euromedservice, Clinical and Diagnostic Center, Moscow
  - MONIKI, Moscow
  - City Clinical Hospital #1 n.a. A.N. Kabanov, Omsk
  - Vvedenskaya hospital, Saint Petersburg
  - Medical Center "Reavita Med SPb", Saint Petersburg
  - FSBEI HE First Pavlov Medical University, Saint Petersburg
  - Medical Association "NEW HOSPITAL", Yekaterinburg
- South Korea (10):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Centerx, Seoul
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University - Shuang-Ho Hospital, Ministry of Health and Welfare, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raghu G, Richeldi L, Fernandez Perez ER, De Salvo MC, Silva RS, Song JW, Ogura T, Xu ZJ, Belloli EA, Zhang X, Seid LL, Poole L; ZEPHYRUS-1 Study Investigators. Pamrevlumab for Idiopathic Pulmonary Fibrosis: The ZEPHYRUS-1 Randomized Clinical Trial. JAMA. 2024 Aug 6;332(5):380-389. doi: 10.1001/jama.2024.8693. PMID 38762797
- [Derived] Rayego-Mateos S, Morgado-Pascual JL, Lavoz C, Rodrigues-Diez RR, Marquez-Exposito L, Tejera-Munoz A, Tejedor-Santamaria L, Rubio-Soto I, Marchant V, Ruiz-Ortega M. CCN2 Binds to Tubular Epithelial Cells in the Kidney. Biomolecules. 2022 Feb 3;12(2):252. doi: 10.3390/biom12020252. PMID 35204752

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a double-blind (DB) period (main study cohort and Japan extension cohort) and an open-label extension (OLE) period. OLE period was not conducted in Japan.
  The efficacy outcome measures data were not collected for Japan cohorts due to early termination of study.
Groups:
- Main Study Cohort: Pamrevlumab: Participants received pamrevlumab 30 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion every 3 weeks for up to 48 weeks in the DB period and continued to receive the same dose of pamrevlumab for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of idiopathic pulmonary fibrosis (IPF), or the sponsor decided to end the OLE period, whichever occurred first.
- Main Study Cohort: Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks in the DB period. Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of IPF, or the sponsor decided to end the OLE period, whichever occurred first.
- Japan Extension Cohort: Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
- Japan Extension Cohort: Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks.
Period: DB Period (48 Weeks)
Arm/Group | Main Study Cohort: Pamrevlumab | Main Study Cohort: Placebo | Japan Extension Cohort: Pamrevlumab | Japan Extension Cohort: Placebo
Started | 181 | 175 | 18 | 19
Received at Least 1 Dose of Study Drug | 181 | 175 | 18 | 19
Completed | 146 | 134 | 14 | 11
Not Completed | 35 | 41 | 4 | 8
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 4
Not completed — Adverse Event | 2 | 5 | 1 | 2
Not completed — Death | 13 | 17 | 1 | 0
Not completed — Investigator Decision | 2 | 2 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 0 | 1
Not completed — Noncompliance with the Study Drug | 1 | 1 | 0 | 0
Not completed — Lung Transplant | 0 | 1 | 0 | 0
Not completed — Participant Decision | 9 | 12 | 1 | 1
Period: OLE (Maximum Exposure: 153.1 Weeks)
Arm/Group | Main Study Cohort: Pamrevlumab | Main Study Cohort: Placebo | Japan Extension Cohort: Pamrevlumab | Japan Extension Cohort: Placebo
Started | 129 (17 participants who completed DB period did not continue in to the OLE period.) | 123 (11 participants who completed DB period did not continue in to the OLE period.) | 0 | 0
Received at Least 1 Dose of Study Drug | 129 | 123 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 129 | 123 | 0 | 0
Not completed — Adverse Event | 7 | 1 | 0 | 0
Not completed — Death | 12 | 12 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Investigator Decision | 2 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 84 | 88 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0 | 0
Not completed — Lung Transplant | 2 | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0
Not completed — Participant Decision | 12 | 13 | 0 | 0
Not completed — Other than specified | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- DB Period (Main Study Cohort): Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the DB period and continued to receive the same dose of pamrevlumab for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of IPF, or the sponsor decided to end the OLE period, whichever occurred first.
- DB Period (Main Study Cohort): Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks in the DB period. Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of IPF, or the sponsor decided to end the OLE period, whichever occurred first.
- DB Period (Japan Extension Cohort): Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
- DB Period (Japan Extension Cohort): Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | DB Period (Main Study Cohort): Pamrevlumab | DB Period (Main Study Cohort): Placebo | DB Period (Japan Extension Cohort): Pamrevlumab | DB Period (Japan Extension Cohort): Placebo | Total
Number analyzed (Participants) | 181 | 175 | 18 | 19 | 393
Age, Customized [Count of Participants; unit: Participants]
  ≤64 Years | 41 | 28 | 3 | 5 | 77
  65 - 74 Years | 77 | 94 | 10 | 5 | 186
  ≥75 Years | 63 | 53 | 5 | 9 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 5 | 3 | 106
  Male | 132 | 126 | 13 | 16 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 44 | 0 | 0 | 98
  Not Hispanic or Latino | 127 | 131 | 18 | 19 | 295
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 63 | 69 | 18 | 19 | 169
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 117 | 104 | 0 | 0 | 221
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] — FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that could forcibly be blown out after full inspiration in the upright position, measured in liters. Population: Per planned analysis, the Baseline characteristics data for 'main study cohort' and 'Japan extension cohort' was collected and reported separately.
  liters
    Main Study Cohort: number analyzed (Participants) | 181 | 175 | 0 | 0 | 356
    Main Study Cohort | 2.3668 (0.6185) | 2.4161 (0.6453) |  |  | 2.3911 (0.6314)
    Japan Extension Cohort: number analyzed (Participants) | 0 | 0 | 18 | 19 | 37
    Japan Extension Cohort |  |  | 2.5864 (0.5521) | 2.5486 (0.5153) | 2.5670 (0.5264)

OUTCOME MEASURES:

1. Primary Outcome: DB Period (Main Study Cohort): Change From Baseline in FVC at Week 48
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that could forcibly be blown out after full inspiration in the upright position, measured in liters. Least square (LS) mean and standard error (SE) were calculated using mixed model for repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- DB Period (Main Study Cohort) - Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
- DB Period (Main Study Cohort) - Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks.
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 163 | 149
liters | -0.26 (0.046) | -0.33 (0.050)
Statistical Analysis 1: Comparison: DB Period (Main Study Cohort) - Pamrevlumab vs DB Period (Main Study Cohort) - Placebo; Test type: Other; p = 0.2926, Mixed Models Analysis; LS Mean Difference = 0.07, 95% CI 2-sided [-0.06 to 0.19], Standard Error of Mean 0.062

2. Primary Outcome: DB Period (Japan Extension Cohort): Change From Baseline in FVC at Week 48
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that could forcibly be blown out after full inspiration in the upright position, measured in liters.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Groups:
- DB Period (Japan Extension Cohort) - Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
- DB Period (Japan Extension Cohort) - Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks.
Arm/Group | DB Period (Japan Extension Cohort) - Pamrevlumab | DB Period (Japan Extension Cohort) - Placebo
Number analyzed (Participants) | 15 | 15
liters | -0.0445 (0.1805) | -0.1835 (0.2389)

3. Secondary Outcome: DB Period (Main Study Cohort): Time to Disease Progression
Description: Time to disease progression was defined as the number of weeks from randomization to either the first occurrence of an absolute ≥10% decline from baseline in percent predicted FVC (FVCpp) or all-cause death, whichever occurred first. Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. Hence, the 'Median Time to Event' is longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 49 | 56
weeks | 54.3 [52.7 to NA] — Due to the low number of participants with an event, the upper limit of 95% confidence interval (CI) could not be calculated. | 50.7 [50.3 to 54.0]

4. Secondary Outcome: DB Period (Main Study Cohort): Time to First Occurrence of Any Component of the Clinical Composite Endpoint
Description: The components of the clinical composite endpoint included acute IPF exacerbation, respiratory hospitalization, or death. Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. Hence, the 'Median Time to Event' is longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 40 | 45
weeks | 62.7 [59.0 to NA] — Due to the low number of participants with an event, the upper limit of 95% CI could not be calculated. | NA [57.9 to NA] — Due to the low number of participants with an event, median and upper limit of 95% CI could not be calculated.

5. Secondary Outcome: DB Period (Main Study Cohort and Japan Extension Cohort): Change From Baseline in Quantitative Lung Fibrosis (QLF) Volume at Week 48
Description: The QLF volume was calculated as QLF = total lung capacity volume multiplied by percentage (%) of quantitative lung fibrosis for fibrosis of the whole lung. LS mean and SE was calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo | DB Period (Japan Extension Cohort): Pamrevlumab | DB Period (Japan Extension Cohort): Placebo
Number analyzed (Participants) | 157 | 143 | 15 | 15
liters | 251.38 (38.010) | 267.96 (38.763) | 45.08 (88.265) | 78.18 (119.300)

6. Secondary Outcome: DB Period (Main Study Cohort): Time to First Acute IPF Exacerbation
Description: Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. Hence, the 'Median Time to Event' is longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 181 | 175
weeks | 62.7 [62.7 to NA] — Due to the low number of participants with an event, the upper limit of 95% CI could not be calculated. | NA [NA to NA] — Due to the low number of participants with an event, median and 95% CI could not be calculated.

7. Secondary Outcome: DB Period (Main Study Cohort): Time to All-Cause Mortality
Description: as for outcome 6
Time Frame: Up to Week 48
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 181 | 175
weeks | NA [60.6 to NA] — Due to the low number of participants with an event, median and upper limit of 95% CI could not be calculated. | NA [60.1 to NA] — Due to the low number of participants with an event, median and upper limit of 95% CI could not be calculated.

8. Secondary Outcome: DB Period (Main Study Cohort): Time to First Respiratory Hospitalizations
Description: as for outcome 6
Time Frame: Up to Week 48
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DB Period (Main Study Cohort) - Pamrevlumab | DB Period (Main Study Cohort) - Placebo
Number analyzed (Participants) | 181 | 175
weeks | 62.7 [59.0 to NA] — Due to the low number of participants with an event, the upper limit of 95% CI could not be calculated. | NA [57.9 to NA] — Due to the low number of participants with an event, median and upper limit of 95% CI could not be calculated.

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 60 days after last dose of study drug (maximum exposure: 51.1 weeks [in main study cohort DB period], 49.1 weeks [in Japan extension cohort DB period], and 153.1 weeks [in OLE period]
Description: The safety analysis set included all participants who received any study drug.
Groups:
- DB Period (Main Study Cohort): Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the DB period.
- DB Period (Main Study Cohort): Placebo: Participants received placebo matched to pamrevlumab by IV infusion every 3 weeks for up to 48 weeks in the DB period.
- DB Period (Japan Extension Cohort)Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks.
- OLE Period: Pamrevlumab/Pamrevlumab: Participants who received pamrevlumab in the DB period continued to receive the same dose of pamrevlumab for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of IPF, or the sponsor decided to end the OLE period, whichever occurred first.
- OLE Period: Placebo/Pamrevlumab: Participants who received placebo matched to pamrevlumab in the DB period, received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for up to 48 weeks in the OLE period or until pamrevlumab was commercially available for the indication of IPF, or the sponsor decided to end the OLE period, whichever occurred first.
Arm/Group | DB Period (Main Study Cohort): Pamrevlumab | DB Period (Main Study Cohort): Placebo | DB Period (Japan Extension Cohort)Pamrevlumab | DB Period (Japan Extension Cohort): Placebo | OLE Period: Pamrevlumab/Pamrevlumab | OLE Period: Placebo/Pamrevlumab
All-Cause Mortality (participants affected / at risk) | 23/181 | 22/175 | 1/18 | 2/19 | 17/129 | 14/123
Serious Adverse Events (participants affected / at risk) | 51/181 | 60/175 | 5/18 | 8/19 | 42/129 | 33/123
Other Adverse Events (participants affected / at risk) | 129/181 | 121/175 | 17/18 | 16/19 | 76/129 | 75/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period (Main Study Cohort): Pamrevlumab (N=181) | DB Period (Main Study Cohort): Placebo (N=175) | DB Period (Japan Extension Cohort)Pamrevlumab (N=18) | DB Period (Japan Extension Cohort): Placebo (N=19) | OLE Period: Pamrevlumab/Pamrevlumab (N=129) | OLE Period: Placebo/Pamrevlumab (N=123)
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 8 | 8 | 1 | 1 | 5 | 4
COVID-19 (Infections and infestations) | 3 | 1 | 0 | 1 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 2 | 3 | 16 | 14
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac perforation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 3 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 5 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Lyme carditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vaccine breakthrough infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 0 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period (Main Study Cohort): Pamrevlumab (N=181) | DB Period (Main Study Cohort): Placebo (N=175) | DB Period (Japan Extension Cohort)Pamrevlumab (N=18) | DB Period (Japan Extension Cohort): Placebo (N=19) | OLE Period: Pamrevlumab/Pamrevlumab (N=129) | OLE Period: Placebo/Pamrevlumab (N=123)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0 | 2 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 3 | 2
Cataract (Eye disorders) | 2 | 0 | 0 | 1 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 1 | 3 | 1
Scleritis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 1 | 2 | 0 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 4 | 4 | 8 | 5
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 7 | 0 | 1 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 0 | 1 | 5 | 2
Oesophageal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0 | 2 | 0 | 1
Chest pain (General disorders) | 3 | 4 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 12 | 10 | 0 | 0 | 8 | 3
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 0 | 1 | 3 | 0
Pyrexia (General disorders) | 1 | 7 | 1 | 2 | 2 | 5
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 14 | 14 | 0 | 0 | 15 | 9
COVID-19 (Infections and infestations) | 22 | 16 | 5 | 2 | 14 | 11
Cystitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 6 | 1 | 3 | 6 | 3
Pneumonia (Infections and infestations) | 6 | 7 | 0 | 1 | 4 | 3
Sinusitis (Infections and infestations) | 4 | 5 | 1 | 0 | 1 | 5
Tinea pedis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 5 | 0 | 1 | 4 | 5
Urinary tract infection (Infections and infestations) | 3 | 3 | 0 | 1 | 5 | 6
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 0 | 1 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 3 | 0 | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 1 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 6 | 11 | 0 | 2 | 3 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 0 | 1 | 5 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1 | 0 | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 1 | 1 | 2 | 4
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 1 | 3 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 10 | 7 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 13 | 12 | 0 | 0 | 3 | 4
Olfactory dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 5 | 2 | 1 | 1 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 25 | 3 | 2 | 11 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 16 | 0 | 0 | 9 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 1 | 7 | 7 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 2 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 2 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 11 | 5 | 0 | 0 | 1 | 3

LIMITATIONS AND CAVEATS:
Study did not meet its primary endpoint; hence, it was terminated early. The Japan extension cohort and OLE period were halted due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT03955146/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03955146/SAP_001.pdf